CLINICAL TRIAL: NCT00060125
Title: PHASE II TRIAL OF R115777 IN PATIENTS WITH METASTATIC MALIGNANT MELANOMA
Brief Title: Tipifarnib in Treating Patients With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02958; CALGB-500104; CDR0000299508; U10CA031946 (NIH)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — tipifarnib

ARMS (1):
- Treatment (tipifarnib) (Experimental): Patients receive oral tipifarnib twice daily on days 1-21. Treatment repeats every 28 days for at least 2 courses and for a maximum of 2 years in the absence of disease progression or unacceptable toxicity. Patients who achieve CR receive 2 additional courses beyond CR.
  Interventions: Drug: tipifarnib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well tipifarnib works in treating patients with metastatic malignant melanoma. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the clinical response rate in patients with metastatic malignant melanoma treated with R115777 (tipifarnib).

II. To evaluate the safety of R115777 in patients with metastatic melanoma.

SECONDARY OBJECTIVES:

I. To assess RhoC expression in tumor samples pre- and post- therapy with R115777.

II. To evaluate Ftase levels in peripheral blood and tumor samples pre- and post-therapy with R115777.

III. To assess the effect of R115777 treatment on T lymphocyte cytokine production, pre- and post- therapy with R115777.

IV. Estimate time to treatment failure (TTF). Time to treatment failure is defined as time to withdrawal for unacceptable toxicity or progressive disease.

OUTLINE Patients receive oral tipifarnib twice daily on days 1-21. Treatment repeats every 28 days for at least 2 courses and for a maximum of 2 years in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (CR) receive 2 additional courses beyond CR.

Patients who discontinue therapy due to toxicity or complete response are followed every 3 months for 2 years after study entry. Patients who discontinue therapy due to disease progression are followed every 6 months for 2 years after study entry. Patients with stable or partially responding disease who complete treatment are followed at 2 years after study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of cutaneous melanoma and clinical evidence of distant metastatic, non-resectable regional lymphatic, or extensive in transit recurrent disease
* Patients must have at least 2 cutaneous lesions amenable to excisional biopsy for correlative studies; in addition, patients must have measurable disease; the disease remaining after the first excisional biopsy must be measurable; lesions that are considered intrinsically non-measurable include the following:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
  * Lesions that are situated in a previously irradiated area
* No history of brain metastases
* No allergies to azoles (e.g. ketoconazole) or allergies to compounds structurally similar to R115777
* No more than 1 prior immunotherapy regimen for treatment of advanced melanoma; an additional immunologic therapy in the adjuvant setting (e.g. IFN-a) is acceptable; prior chemotherapy for any stage of melanoma is not allowed

  * No radiotherapy or immunotherapy within four weeks prior to the initiation of therapy on this study
* CTC (ECOG) performance status 0-1
* Non-pregnant, non-nursing; treatment under this protocol would expose an unborn child to significant risks; women and men of reproductive potential should agree to use an effective means of birth control; women of child-bearing age will undergo pregnancy testing
* ANC >= 1500/uL
* Platelets >= 100,000/uL
* Bilirubin =< 1.5 mg/dL
* Creatinine =< 2.0 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-05; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Response rate (complete response [CR] and partial response [PR]} | Up to 2 years
  Estimated confidence intervals will be adjusted for the number of stages.
Progression-free survival (PFS) | From date of entry onto the trial until documented progression or death from any cause, assessed up to 2 years
  Estimated using the method of Kaplan and Meier.
Time to treatment failure (TTF) | From trial entry until a patient ends protocol therapy due to unacceptable toxicity, progression or death from any cause, assessed up to 2 years
  Estimated using the method of Kaplan and Meier.

SECONDARY OUTCOMES:
Correlation between RhoC expression levels and response | From baseline to up to 2 years
Change in FTAse levels | From baseline to up to 2 years
Change in the production of IL-2 and IFN-g by T cells | From baseline to up to 2 years
  Descriptive statistics will be used to describe the mean and spread of production of IL-2 and IFN-g.
Adverse events as assessed by Common Toxicity Criteria (CTC) version 2.0 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gajewski, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States

REFERENCES:
- [Derived] Gajewski TF, Salama AK, Niedzwiecki D, Johnson J, Linette G, Bucher C, Blaskovich MA, Sebti SM, Haluska F; Cancer and Leukemia Group B. Phase II study of the farnesyltransferase inhibitor R115777 in advanced melanoma (CALGB 500104). J Transl Med. 2012 Dec 10;10:246. doi: 10.1186/1479-5876-10-246. PMID 23228035